CLINICAL TRIAL: NCT05104606
Title: Speckle Tracking Evaluation of the Impact of Inhaled Nitric Oxide on the Right Ventricle in Acute Respiratory Distress Syndrome
Brief Title: Speckle Tracking and Inhaled Nitric Oxide in Acute Respiratory Distress Syndrome
Acronym: NOSPECKLE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PI2021_843_0066
Record Dates: First submitted 2021-10-12; First posted 2021-11-03 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: ARDS; Right Ventricle
Keywords: speckle tracking; ARDS; right ventricle; iNO; strain
MeSH Terms: conditions — Sprains and Strains

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: TEE — The intervention within the framework of the protocol will consist, for the needs of the study, in performing 2 TEE and 5 TTE in 24 hours after
  For TEE:
  * The first TEE will allow us to evaluate the right ventricle, to look for the existence of a acute cor pulmonale, to evaluate the patient's blood volume as recommended during the management of ARDS. If the patient is included in the study, our intervention will consist in leaving this TEE in place in order to perform measurements at H0, 30min, H1 and H2 after iNO administration.
  * The second TEE will be performed at H24 to performed new measurements.
Other: TTE — For TTE:
  • The TTEs will allow us to evaluate the anatomy of the right ventricle, to estimate the systolic pulmonary artery pressure, to calculate the cardiac output and to measure the conventional parameters of the right ventricular systolic function. This noninvasive examination will be repeated at 30 min, H1, H2, and H24 after iNO administration

SUMMARY:
Acute cor pulmonale is one of deadly complications of mechanically ventilated acute respiratory distress syndrome (ARDS), which can lead to right ventricular dysfunction and worsen the hemodynamics of the patient. For several years, transthoracic (TTE) and transesophageal echocardiography (TEE) have replaced the pulmonary artery catheter to monitor cardiac function reliably and non-invasively.

Speckle tracking is an echocardiographic technique that allows a two-dimensional strain (2D) analysis of right ventricular systolic function. Right ventricular global strain (RVGLS) is a strain parameter, allowing an early and more accurate diagnosis of right ventricular dysfunction than conventional parameters.

This project will consist of performing TTE and TEE measurements at H0, 30min, H1, H2, and H24 after iNO administration in patient with ARDS under mechanical ventilation. The patient will be declared responder to iNO, if there is an increase of more than 20% of the PaO2/FiO2. 30 minutes after a dose of 10ppm of iNO.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (age > 18 years)
* Hospitalized in the intensive care and post-operative care unit of the Amiens-Picardie University Hospital
* Patient with ARDS (defined by the Berlin criteria) requiring mechanical ventilation with a P/F ratio < 200 and requiring iNO
* Beneficiary of social security
* Signature of the consent to participate in the study by the patient or, if unconscious, his legal representative/next of kin

Exclusion Criteria:

* Pregnant or breastfeeding woman
* Contraindications to TEE (major upper gastro-intestinal surgery, mediastinal radiotherapy, active esophagitis, esophageal varices)
* Contraindications to the placement of an esophageal probe (recent upper gastro-intestinal surgery, active ulcer, active esophagitis)
* Presence of atrial fibrillation on echocardiographic examinations
* Contraindications to the administration of iNO
* Patients with chronic treatment allowing pulmonary arterial vasodilatation by sildenafil.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2021-11-02 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Variation from baseline of systolic function after iNO administration | 30 minutes
  Systolic function will be assessed with "in speckle tracking RV" in the presence or not of a response to iNO 30 minutes after its administration, Systolic function will be assessed with "in speckle tracking RV" in patients with moderate to severe ARDS under mechanical ventilation.

SECONDARY OUTCOMES:
Variation from baseline of systolic function after iNO administration | at 1 hour
  Right ventricular function is assessed by speckle tracking at 1 hour after iNO administration in iNO responders
Variation from baseline of systolic function after iNO administration | at 1 hour
  Right ventricular function is assessed by speckle tracking at 1 hour after iNO administration in iNO nonresponders
Variation from baseline of systolic function after iNO administration | at 2 hours
  Right ventricular function is assessed by speckle tracking at 2 hours after iNO administration in iNO responders
Variation from baseline of systolic function after iNO administration | at 2 hours
  Right ventricular function is assessed by speckle tracking at 2 hours after iNO administration in iNO nonresponders
Variation from baseline of systolic function after iNO administration | at 24 hours
  Right ventricular function is assessed by speckle tracking at 24 hours after iNO administration in iNO responders
Variation from baseline of systolic function after iNO administration | at 24 hours
  Right ventricular function is assessed by speckle tracking at 24 hours after iNO administration in iNO nonresponders

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens Picardie, Amiens, France

IPD SHARING:
Plan to Share IPD: No